CLINICAL TRIAL: NCT05587816
Title: Evaluating the Validity of a Novel Tool to Measure Children's Food Intake and Improve Health
Brief Title: Validity of the PortionSize App to Measure Children's Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Blue Cross and Blue Shield of Louisiana Foundation (Unknown)
Responsible Party: Principal Investigator, Hanim Diktas, Principal Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBRC 2022-031
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Nutritional Assessment
Keywords: Dietary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): * Training and use of the PortionSize app by children and parents or caregivers
  * Using the PortionSize app at the clinic of Pennington Biomedical Research Center and at home (free-living condition)
  * Rating the satisfaction of using the PortionSize app
  Interventions: Device: Validation of the PortionSize app

INTERVENTIONS:
Device: Validation of the PortionSize app — The investigators will recruit 40 dyads (40 children aged 7-12 years old and 40 parents or caregivers) using a convenience sample for this pilot study. Children and their parents or caregivers will be trained to use the PortionSize app at Pennington Biomedical Research Center (PBRC). Children will use the PortionSize app and estimate food intake from pre-weighed meals (simulated meals) at PBRC clinic. Children will not consume the simulated meals. Children's parents or caregivers will also use the PortionSize app and estimate the food intake of their children (at least one meal and a snack each day) for two consecutive days at home.

SUMMARY:
The purpose of this study is to assess the validity of the PortionSize™ app to quantify children's own dietary intake and children's intake by parents or caregivers.

DETAILED DESCRIPTION:
The investigators will recruit 40 dyads (40 children aged 7-12 years old and 40 parents or caregivers) using a convenience sample for this pilot study. Children and their parents or caregivers will be trained to use the PortionSize app at Pennington Biomedical Research Center (PBRC). Children will use the PortionSize app and estimate food intake from pre-weighed meals (simulated meals) at PBRC clinic. Children will not consume the simulated meals. Children's parents or caregivers will also use the PortionSize app and estimate the food intake of their children (at least one meal and a snack each day) for two consecutive days at home.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Children (7-12 years) and their parents or caregivers (18-62 years)
* Parents who have Willingness to use the PortionSize app to estimate the intake of their child food intake (normal/regular diet) from at least a snack and a meal of child for two consecutive days
* Have iPhone (version 6 or above) and an operable Apple ID, password, and email address, and able to use iPhone

Exclusion Criteria:

* Any condition or circumstance that could impede study completion
* Child who is a very choosy eater or has a very limited food choice

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Estimation of energy intake (kcal) by children using the PortionSize app | One study visit of ~ 2.5 hours
  Percent mean error and Bland-Altman analysis will be performed to determine errors in estimations of energy intake from the PortionSize app compared to estimations of energy intake from the weighed meals (the criterion measure).
Estimation of intake of food group servings (fruit, vegetable, grain, protein, and dairy) by children using the PortionSize app | One study visit of ~ 2.5 hours
  Percent mean error and Bland-Altman analysis will be performed to determine errors in estimations of intake of food group servings from the PortionSize app compared to estimations of food group servings from the weighed meals (the criterion measure).
Estimation of energy intake (kcal) by parents or caregivers using the PortionSize app | Parents or caregivers will assess food intake of their child (at least one meal and a snack) for two consecutive days at home
  Percent mean error and Bland-Altman analysis will be performed to assess errors in estimating energy intake using the PortionSize app compared to estimations of energy measured by expert raters via food photography analysis.
Estimation of intake of food group servings (fruit, vegetable, grain, protein, and dairy) by parents or caregivers using the PortionSize app | Parents or caregivers will assess food intake of their child (at least one meal and a snack) for two consecutive days at home
  Percent mean error and Bland-Altman analysis will be performed to assess errors in intake of food group servings using the PortionSize app compared to estimations of food group servings measured by expert raters via food photography analysis.

SECONDARY OUTCOMES:
User satisfaction of the PortionSize app for recording food intake by children | One study visit of ~ 2.5 hours
  After completing assessment of food at clinic, children will complete a Likert scale-based survey questionnaire (User Satisfaction questionnaire). The investigators updated a 10-question user satisfaction survey that has been administered in prior studies to quantify satisfaction, ease of use, and adequacy of training for mobile app. The minimum value is 1 and the maximum value is 6 for each question and higher scores indicate a higher outcome.
User satisfaction of the PortionSize app for recording food intake by parents or caregivers | Parents or caregivers will assess food intake of their child (at least one meal and a snack) for two consecutive days at home
  After completing assessment of child's food intake, parents or caregivers will complete a Likert scale-based survey questionnaire (User Satisfaction questionnaire). . The investigators updated a 10-question user satisfaction survey that has been administered in prior studies to quantify satisfaction, ease of use, and adequacy of training for mobile app. The minimum value is 1 and the maximum value is 6 for each question and higher scores indicate a higher outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hanim E Diktas, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Any identifiers might be removed from the participants identifiable information and after the removal, the information could be used for future research studies or given to another investigator for future research without additional informed consent from the subject or legally authorized representative.